CLINICAL TRIAL: NCT02219191
Title: The Effect of Puerarin Tablets in Treating Metabolism Syndrome in Patients With Chronic Rheumatic Diseases
Brief Title: Puerarin Versus Atorvastatin in Treating Metabolism Syndrome in Patients With Chronic Rheumatic Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chengdu PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yang Min, Ph.D, Chengdu PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTSTA20141102
Record Dates: First submitted 2014-07-16; First posted 2014-08-18 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Puerarin tablet; rheumatoid arthritis; metabolism syndrome
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — puerarin; Atorvastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- puerarin tablet 50 mg (Experimental): Patients were orally administrated with 50 mg puerarin tablet three times a day for 24 weeks. Furthermore, patients receive stable treatment with oral anti-rheumatic agents and/or non-steroidal anti-inflammatory drugs, prednisone, aspirin, bone metabolism regulators and gastric mucosal protective agents on as-needed basis.
  Interventions: Drug: puerarin tablet 50 mg
- Atorvastatin tablet 20 mg (Active Comparator): Patients were orally administrated with 20 mg Atorvastatin tablet once a day for 24 weeks. Furthermore, patients receive stable treatment with oral anti-rheumatic agents and/or non-steroidal anti-inflammatory drugs, prednisone, aspirin, bone metabolism regulators and gastric mucosal protective agents on as-needed basis.
  Interventions: Drug: Atorvastatin tablet 20 mg

INTERVENTIONS:
Drug: puerarin tablet 50 mg
  Other Names: C15H10O4254.24
  Arms: puerarin tablet 50 mg
Drug: Atorvastatin tablet 20 mg — Approval No.: H19990258
  Other Names: (3r,5rr)-7-[2-(4-fluorophenyl)-3-phenyl-4-(phenylcarbamoyl)-5-propan-2-yl-pyrrol-1-yl]-3,5-dihydroxy-heptanoic acid
  Arms: Atorvastatin tablet 20 mg

SUMMARY:
To evaluate the Effect of Puerarin tablets versus statins in treating metabolism syndrome in patients with chronic rheumatic diseases

ELIGIBILITY:
Inclusion Criteria:

* patients with a definite diagnose with rheumatic disease
* patients with metabolic Syndrome
* without conflict to the written, informed consent signed prior to the enrollment
* no severe hepatic or renal disorders
* no known carotid artery stenosis
* no coagulation disorders
* no hypertension

Exclusion Criteria:

* being in pregnancy, lactation period or under a pregnancy plan
* being allergic to the test drug
* not compatible for the trial medication
* without full legal capacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in homeostasis model assessment (HOMA-IR) | At 0 week, 12 weeks, 24 weeks and 48 weeks

SECONDARY OUTCOMES:
Fasting serum low-density lipoprotein cholesterol (LDL-C) | at 0 week, 12 weeks, 24 weeks, 48 weeks
Fasting serum high-density lipoprotein cholesterol (HDL-C) | at 0 week, 12 weeks, 24 weeks, 48 weeks
erythrocyte sedimentation rate (ESR) | at 0 week, 12 weeks, 24 weeks, 48 weeks
C reactive protein (CRP) | at 0 week, 12 weeks, 24 weeks, 48 weeks
Fasting serum total cholesterol (TC) | at 0 week, 12 weeks, 24 weeks, 48 weeks
Fasting serum triglycerides (TGs) | at 0 week, 12 weeks, 24 weeks, 48 weeks
tumor necrosis factor (TNFα) | at 0 week, 12 weeks, 24 weeks, 48 weeks
interleukin-8 (IL-8) | at 0 week, 12 weeks, 24 weeks, 48 weeks
interleukin-1 (IL-1) | at 0 week, 12 weeks, 24 weeks, 48 weeks
interleukin-6 (IL-6) | at 0 week, 12 weeks, 24 weeks, 48 weeks
Fasting serum insulin | at 0 week, 12 weeks, 24 weeks, 48 weeks
Fasting serum glucose | at 0 week, 12 weeks, 24 weeks, 48 weeks
Kidney function | at 0 week, 12 weeks, 24 weeks, 48 weeks
Liver function | at 0 week, 12 weeks, 24 weeks, 48 weeks
blood cell count | at 0 week, 12 weeks, 24 weeks, 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- 270 Rongdu street, Jin-niu district,Rheumatology Center of Integrated Medicine, General Hospital of Chengdu Military Area Command PLA，, Chengdu, Sichuan, China